CLINICAL TRIAL: NCT01450020
Title: Sister Survivor: Improving the Survivorship Care of African-American Women With Breast Cancer
Brief Title: Peer Navigator Education in Improving Survivorship Care in African American Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11115; NCI-2011-03229 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: cancer survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Methods; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (PN and ACS material) (Experimental): Participants receive 4 PN sessions tailored to their needs followed by a 6 month booster session and ACS materials.
  Interventions: Other: educational intervention; Other: questionnaire administration; Other: counseling intervention; Other: survey administration; Procedure: quality-of-life assessment
- Arm II (ACS material) (Active Comparator): Participants receive ACS materials only.
  Interventions: Other: educational intervention; Other: questionnaire administration; Other: survey administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Receive ACS material
  Other Names: intervention, educational
Other: questionnaire administration — Ancillary studies
Other: counseling intervention — Undergo PN session
  Other Names: counseling and communications studies
  Arms: Arm I (PN and ACS material)
Other: survey administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized clinical trial studies peer navigator education in improving survivorship care in African American breast cancer survivors. An educational intervention involving peer groups may help to improve the well-being and quality of life (QOL) in breast cancer survivors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the ability of peer navigation (PN) to improve understanding of survivorship care planning (SCP) at 6 months.

II. To promote adherence to the SCP schedule of follow-up examinations at 12 months.

SECONDARY OBJECTIVES:

I. To evaluate the effect of PN on change from baseline in medical efficacy, preparedness for life as new survivor, and physical and health related QOL at 6 months.

OUTLINE: PNs are trained on medical issues and resources, and SCP. Participants are then randomized to 1 of 2 treatment arms.

ARM I: Participants receive 4 PN sessions tailored to their needs followed by a 6 month booster session and American Cancer Society (ACS) materials.

ARM II: Participants receive ACS materials.

After completion of study treatment, patients are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* TRIAL SUBJECTS:
* Patient age 18 years or older who self-identifies as African-American
* In early survivorship phase, defined as being 1-12 months post completion of treatment for stage 0-3 breast cancer
* Receiving health care primarily through an health maintenance organization (HMO)
* Patients with metastatic cancer or a second primary cancer, because their medical characteristics (e.g. disease progression) are significantly different
* Breast cancer survivors (BCS) with other major disabling medical, psychiatric, or substance abuse conditions (e.g., anxiety, depression, alcohol/tobacco problems) will be excluded
* PEER NAVIGATORS:
* At least 25 years of age who self-identifies as African-American
* Previously participated in any type of research study
* Has at least high school education
* Has been diagnosed with breast cancer, currently in remission or eradicated
* Belongs to a breast cancer support group
* Has a valid driver's license
* Owns an operational vehicle
* Has access to a personal computer with internet access

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2012-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ability of peer navigation to improve understanding of SCP | At 6 months
  Chi-square and t-tests will be used to compare the baseline characteristics of subjects randomized to PN intervention vs control. For subjects in the intervention arm, the number of navigation sessions received will be reported, and correlated factors will be explored. The number of subjects navigated per PN will also be reported. Nonevaluable and evaluable subjects (defined at 6 and 12 months) will be compared. Site of care will be handled as a cluster level variable in generalized linear mixed (GLM) regression models.
Adherence to the SCP schedule of follow-up examinations | At 12 months
  Measured using a newly created, 50-point scale that gives equal weight to completion of the recommended: physical exams, imaging, pelvic exam, annual oncology visit, and breast self-exams.

SECONDARY OUTCOMES:
Effect of PN on change in medical efficacy | Baseline to 6 months
  Exploratory analyses will analyze the effect of PN intervention actually received, using the number of PN sessions completed and the quality of the subject's PN as measured by PN's post-training level of acuity and utility.
Preparedness for life as new survivor (PLANS) | At 6 months
  PLANS consists of two subscales that measure patients' knowledge and self efficacy with regards to their Access and Quality of Survivorship Care Plan (SCP) and adherence with regard to following these tasks. The knowledge subscale (Cronbach's alpha 0.90) and adherence subscale (Cronbach's alpha 0.70) have good reliability.
Physical and health related QOL | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States